CLINICAL TRIAL: NCT04144543
Title: Experimental Randomized Study: The Effect of White Noise and Facilitated Tucking Applications During Heel-Stick Sampling on Pain in Term Babies
Brief Title: Non-pharmacological Pain Management in Term Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Aylin PEKYİGİT, Research Assistant, Çankırı Karatekin University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Eskisehir Osmangazi University
Record Dates: First submitted 2019-10-23; First posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Facilitated Tucking

STUDY DESIGN:
Intervention Model Description: White Noise Group:
  The white noise was initiated 50 cm away from the baby, with the decibel meter set to an average of 55 decibels. The baby was exposed to white noise for 2 minutes before the procedure.
  Facilitated Tucking Group:
  The baby's arms and legs were held in flexed positions close to the midline of the torso in side-lying position, so the baby was able to move his/her extremities. The baby was held in facilitated tucking position for one minute before the procedure.
  White Noise+Facilitated Tucking Group:
  The baby was exposed to white noise for 1 minute before the procedure. The white noise was initiated 50 cm away from the baby, with the decibel meter set to an average of 55 decibels. At the second minute, when the white noise still continued to play, facilitated tucking was performed at the same time and the baby continued to listen to the white noise for 1 minute while in facilitated tucking position.
Who Masked: Care Provider, Investigator
Masking Description: Pain scores of the babies before, during and after the procedure were evaluated independently by the researcher and the nurse other than the one who performed heel-stick sampling. Cohen's Kappa test was performed in the evaluation of the NIPS pain scores to test the concordance of the scores given to the same situation by 1 nurse and 1 researcher and it was found that the concordance of the scores given by 2 nurses was perfectly concordant (almost completely concordant) (Kappa Coefficient=0.953, p=0.027).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- White Noise (Experimental): The "white noise" used in our study is a fragment called "Bebeğiniz ağlamasın-2" from "Kolik" album of Buzuki Orhan Osman, which was used in similar studies (Balci, 2006; Karakoc & Turker, 2014; Kucukoglu et al., 2016).Since the white noise is a continuously monotonous sound, which is in the form of a hum, it resembles the sounds in mother's womb (Balci, 2006).
  Interventions: Other: White Noise
- Facilitated Tucking (Experimental): Facilitated tucking is the procedure of holding the baby's arms and legs in a flexed position close to the midline of the torso, and the baby is able to move his/her extremities during this procedure (Caglayan, 2011).
  Interventions: Other: Facilitated Tucking
- White Noise+Facilitated Tucking (Experimental): Both applications performed together.
  Interventions: Other: White Noise+Facilitated Tucking

INTERVENTIONS:
Other: White Noise — The white noise was initiated 50 cm away from the baby, with the decibel meter set to an average of 55 decibels. The baby was exposed to white noise for 2 minutes before the procedure.
  Arms: White Noise
Other: Facilitated Tucking — The baby's arms and legs were held in flexed positions close to the midline of the torso in sidelying position, so the baby was able to move his/her extremities. The baby was held in facilitated tucking position for one minute before the procedure.
  Arms: Facilitated Tucking
Other: White Noise+Facilitated Tucking — The baby was exposed to white noise for 1 minute before the procedure. The white noise was initiated 50 cm away from the baby, with the decibel meter set to an average of 55 decibels. At the second minute, when the white noise still continued to play, facilitated tucking was performed at the same time and the baby continued to listen to the white noise for 1 minute while in facilitated tucking position.
  Arms: White Noise+Facilitated Tucking

SUMMARY:
A randomised clinical trial in a single centre. This study was performed to compare the effect of white noise, facilitated tucking, and their concerted application during heel-stick sampling on pain in term babies.

The study was conducted on 90 babies. Using stratification and blocking method, 30 babies were included in the white noise group (1st Group), 30 in facilitated tucking group (2nd Group), and 30 in white noise + facilitated tucking group (3rd Group). Pain scores of the babies in all groups before, during, and after the procedure were evaluated by two nurses independent from each other using Neonatal Infant Pain Scale (NIPS).

DETAILED DESCRIPTION:
Aims and objectives: This study was performed to compare the effect of white noise, facilitated tucking, and their concerted application during heel-stick sampling on pain in term babies.

Design: A randomised clinical trial in a single centre. Methods: The study sample size was determined by the free-software G* Power. Based on the power analysis performed prior to the study in order to determine the number of babies to be included in the sample group (with β=0.14087 and α=0.05 risk, Power=0.85913), according to the study by Karakoc and Turker (2014), it was found that 27 neonates should be included in each group. The study was conducted on 90 babies, between July 1, 2017 - August 9, 2017. Using stratification and blocking method, 30 babies were included in the white noise group (1st Group), 30 in facilitated tucking group (2nd Group), and 30 in white noise + facilitated tucking group (3rd Group). Pain scores of the babies in all groups before, during, and after the procedure were evaluated by two nurses independent from each other using Neonatal Infant Pain Scale (NIPS).

ELIGIBILITY:
Inclusion Criteria:

* Being term baby
* Being with mother
* Being a healthy baby
* Being able fed orally
* Being fed at least half an hour before the procedure
* Being able to draw blood at the first try (since the pain level will change on the second try)
* Agreed to participate in the study and gave verbal consent were included in the study.

Exclusion Criteria:

* Having received analgesics and/or sedatives within the last 24 hours
* Having any complications that prevent pain evaluation (e.g. intracranial hemorrhage, neuromotor growth retardation, etc.)
* Having undergone any painful procedures within the last hour (e.g. blood drawing, aspiration, ophthalmologic examination, etc.)
* Prior history of surgery
* Being connected to mechanical ventilator

Max Age: 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 90 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-08-09 (Actual); Study Completion 2017-11-24 (Actual)

PRIMARY OUTCOMES:
Pain severity (scores) | 2 MONTHS
  Pain was evaluated separately by NIPS by two individuals, one investigator and one nursing nurse. The scores given by the investigator and the nurse were used to determine pain scores before, during and after heel blood collection. Pain severity was expressed as mean score NIPS.Neonatal Infant Pain Scale (NIPS) was used in the evaluation of the pain of the neonates. This scale was developed by Lawrence et al. (1993). The validity and reliability of the Turkish version of the test were assessed by Akdovan (1999). There are six variables in the scale. These are baby's breathing pattern, wakefulness, crying, facial movements and arm and leg movements. These variables are scored between 0-1. Only crying is scored between 0-2. The total score is between 0-7. The resulting score is directly proportional to the severity of the pain. That is, as the score increases, the severity of the pain increases (Akdovan, 1999). The study was completed with 90 infants.

SECONDARY OUTCOMES:
Crying time | 2 MONTHS
  The researcher recorded the crying time in second (sec) during and after heel blood collection. The study was completed with 90 infants.

OTHER OUTCOMES:
Physiological Changes: Heart rate | 2 MONTHS
  The pulse oximetry probe was attached to a non-heeled foot to measure heart in second (sec) before, during and after heel blood collection in each infant. The study was completed with 90 infants.
Physiological Changes: Oxygen saturation | 2 MONTHS
  The pulse oximetry probe was attached to a non-heeled foot to measure oxygen saturation in percent (%) before, during and after heel blood collection in each infant. The study was completed with 90 infants.
Physiological Changes: Respiration | 2 MONTHS
  The researcher recorded the respiration in minute (min) before and after heel blood collection. The study was completed with 90 infants.

CONTACTS AND LOCATIONS:
Locations (1):
- Çankırı Karatekin Üniversitesi, Çankiri, Turkey (Türkiye)

REFERENCES:
- [Background] Karakoc A, Turker F. Effects of white noise and holding on pain perception in newborns. Pain Manag Nurs. 2014 Dec;15(4):864-70. doi: 10.1016/j.pmn.2014.01.002. Epub 2014 Feb 20. PMID 24559599
- [Background] Kucukoglu S, Aytekin A, Celebioglu A, Celebi A, Caner I, Maden R. Effect of White Noise in Relieving Vaccination Pain in Premature Infants. Pain Manag Nurs. 2016 Dec;17(6):392-400. doi: 10.1016/j.pmn.2016.08.006. Epub 2016 Oct 15. PMID 27751753
- [Background] Caglayan, N. (2011). The effect on pain of manipulating the preterm neonate into the facilitated tucking during drawing of blood from the heel. Turkey: Unpublished Master Thesis. Istanbul University Health Sciences Institute, Istanbul. Retrived from https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp
- [Background] Balci, S. (2006). Effect of white noise in colicky baby. Turkey: Unpublished Master's Thesis, Marmara University Institute of Health Sciences, Istanbul. Retrived from: https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp
- [Background] Akdovan, T. (1999). Assessment of pain in healthy newborns, investigation of the effect of the sucking and holding method. Turkey: Unpublisched Master's Dissertation. Marmara University Institute of Health Sciences, Istanbul. Retrived from: https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp
- [Background] Lawrence J, Alcock D, McGrath P, Kay J, MacMurray SB, Dulberg C. The development of a tool to assess neonatal pain. Neonatal Netw. 1993 Sep;12(6):59-66. PMID 8413140